CLINICAL TRIAL: NCT00734513
Title: Partner Assisted Emotional Disclosure for GI Cancer
Brief Title: Partner-Assisted Emotional Disclosure for GI Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00011905; 1R01CA10073-01A1
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2008-08

CONDITIONS: Cancer of the GI System-stages II III and IV
Keywords: GI Cancer; Emotional Disclosure; Behavioral Intervention; Partner; Couples
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Partner-assisted Emotional Disclosure
  Interventions: Behavioral: Partner-assisted emotional disclosure
- 2 (Active Comparator): Cancer Education
  Interventions: Behavioral: Cancer Education

INTERVENTIONS:
Behavioral: Partner-assisted emotional disclosure — Patients and partners in the partner-assisted emotional disclosure condition will attend four weekly face-to-face sessions with a therapist. The first session will last 75 minutes and will focus on training in skills to facilitate the patient's disclosure. The subsequent 3 sessions will last 45 minutes each. In these sessions, the therapist will briefly review the strategies and provide feedback from the previous session and the patient will spend 30 minutes talking about their cancer-related concerns to the partner.
  Other Names: Emotional Disclosure
  Arms: 1
Behavioral: Cancer Education — The cancer education protocol consists of four weekly face-to-face sessions for education about living with GI cancer. The cancer education sessions will be delivered to patients and their partners and use a presentation and discussion format. Handouts and discussion sessions will center on the following topics: Orientation to Duke Cancer Care and the treatment team; suggestions for communicating with health care providers; resources for health information, psychosocial support, and financial concerns; evaluating health information on the internet; the impact of cancer on different domains of quality of life; and suggestions for maintaining quality of life.
  Other Names: Education
  Arms: 2

SUMMARY:
The long-range goal of this research is to develop better ways of helping GI cancer patients and their caregivers cope more effectively with the demands of the disease. The study is designed to test the hypothesis that a partner-assisted emotional disclosure intervention will be more effective in enhancing patient' psychological adjustment than a cancer education condition.

DETAILED DESCRIPTION:
The diagnosis and treatment of GI cancer is a traumatic and life-altering event. Many patients with GI cancer experience significant emotional distress and disruptions in their social relationships as well as multiple physical symptoms and limitations in physical activities. There is evidence that cancer patients who are able to confide their feelings and concerns about the cancer experience with supportive others, particularly their partners, fare better. patients who are able to discuss cancer openly with their partners report fewer emotional and physical complaints, and higher levels of self-esteem and perceived control. However, there are a number of barriers that often inhibit discussion of cancer-related feelings. The proposed study will examine the effect of a new partner-assisted emotional disclosure (ED) protocol for patients with GI cancer.

In this study, 200 patients diagnosed with GI cancer and their partners will be recruited to participate. The couples will be randomly assigned to one of two conditions: 1) partner-assisted emotional disclosure, or 2) cancer education. Assessment measures will be collected at evaluations conducted before and after treatment and at 8 weeks post treatment. All evaluations will be conducted over the phone. Information will also be collected from the physician and/or the patient's medical record at each of the three evaluations. Audiotapes of the partner-assisted emotional disclosure sessions will be transcribed and 10-minute segments will be randomly selected and analyzed to assess the extent to which patients express emotions and partners verbally reflect the partner's feeling in an empathic manner.

ELIGIBILITY:
Inclusion Criteria:

* cancer of the GI system (esophagus, stomach, pancreas, liver, or colorectal; Stage II, III or IV), a life-expectancy of at least 6 months, living with a spouse or intimate partner in a committed relationship, English speaking, and an identified medical oncologist.

Exclusion Criteria:

* None other than absence of inclusion criteria specified above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Patient's psychological adjustment | Immediately after treatment and 8 weeks after completion of treatment

SECONDARY OUTCOMES:
Patient's physical and functional well-being | Immediately after treatment and 8 weeks after completion of treatment
Communication quality between the patient and partner (i.e.level of disclosure, helpfulness of disclosure, and perceived empathy from the partner, and decreased partner avoidance and criticism). | Immediately after treatment and 8 weeks after completion of treatment
Partners' psychological well-being and caregiver strain | Immediately after treatment and 8 weeks after completion of treatment
Gender and marital satisfaction as moderators of the effects of partner-assisted ED. | Immediately after treatment and 8 weeks after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Porter, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States